CLINICAL TRIAL: NCT00693472
Title: Efficacy of SCH 420814 to Reduce the Frequency or Severity of Neuroleptic Induced Akathisia
Brief Title: Study of Preladenant for the Treatment of Neuroleptic Induced Akathisia (Study P05145)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05145; MK-3814-019 (Other: Merck protocol number)
Record Dates: First submitted 2008-05-27; First posted 2008-06-09 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Akathisia, Drug-Induced; Antipsychotic Agents; Movement Disorders
Keywords: Antipsychotic Agents
MeSH Terms: conditions — Akathisia, Drug-Induced; Movement Disorders | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine; Cholinergic Antagonists; Propranolol; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1: Preladenant (Experimental): Preladenant 25 mg every 12 hours for 13 days
  Interventions: Drug: Preladenant; Drug: Anticholinergic agents or propanolol; Drug: Haloperidol
- Part 1: Placebo (Placebo Comparator): Placebo every 12 hours for 13 days
  Interventions: Drug: Placebo; Drug: Anticholinergic agents or propanolol; Drug: Haloperidol
- Part 2: Preladenant (Experimental): Preladenant 25 mg every 12 hours for 13 days
  Interventions: Drug: Preladenant; Drug: Haloperidol
- Part 2: Standard of Care (Active Comparator): Anticholinergic agents or Propranolol as standard-of-care dosing regimen (supplied by the study site)
  Interventions: Drug: Anticholinergic agents or propanolol; Drug: Haloperidol

INTERVENTIONS:
Drug: Preladenant — Preladenant, one 25 mg capsule, administered orally every 12 hours
  Other Names: SCH 420814
  Arms: Part 1: Preladenant; Part 2: Preladenant
Drug: Placebo — Matching placebo capsule administered orally every 12 hours
  Arms: Part 1: Placebo
Drug: Anticholinergic agents or propanolol — Part 1 (as rescue therapy only): participants who develop akathisias may be treated with either anticholinergic agents or propranolol as a rescue medication at the discretion of the treating physician. Individual anticholinergic agents were not pre-specified per protocol.
  Part 2 (standard of care): anticholinergic agents or propanolol at a dose determined by the investigator according to the local standard of care. Individual anticholinergic agents were not pre-specified per protocol.
  Arms: Part 1: Placebo; Part 1: Preladenant; Part 2: Standard of Care
Drug: Haloperidol — Participants continued pre-study haloperidol, admistered orally, at a dose of at least 7.5 mg/day

SUMMARY:
This study is designed to evaluate the effectiveness of preladenant in the prevention (Part 1) or treatment (Part 2) of antipsychotic induced akathisia in participants with acute psychosis using the Barnes Akathisia Scale.

ELIGIBILITY:
Inclusion Criteria:

* Participants or guardian must be willing to give written informed consent.
* Part 1 Only: Participants with acute (not drug related) psychoses with a Positive and Negative Symptom Scale for Schizophrenia (PANSS) score of at least 60: schizophrenia, schizo-affective, schizo-manic, and acute mania with a history of previous treatment with neuroleptics.
* Part 1 Only: Participants initiating haloperidol for the treatment of an acute psychotic episode at a dose of at least 7.5 mg per day.
* Part 2 Only: Inpatient participants who have developed akathisia as a result of haloperidol at >=5 mg per day for the treatment of acute psychosis. The enrollment of participants receiving other neuroleptics is allowed only after consultation and agreement by the sponsor.
* Participants of either sex and of any race between the ages of 18 and 65 years, inclusive.
* Participant's clinical laboratory tests (complete blood count [CBC], blood chemistry, and urinalysis) must be within normal limits or clinically acceptable to the investigator/sponsor. Participant's liver function test results (ie, aspartate aminotransferase [AST], alanine aminotransferase [ALT]) must not be elevated above the normal limits at Screening and on Day -1/1.
* Participants must be free of any clinically significant disease other than psychosis that would interfere with the study evaluations.
* Screening electrocardiogram (ECG) must be clinically acceptable to the investigator.
* Female of childbearing potential must:

  * Have used a medically accepted method of contraception for 1 month (or abstained from sexual intercourse) prior to the screening period. An acceptable method of contraception includes one of the following:

    * condom (male or female) used with spermicide,
    * diaphragm or cervical cap used with spermicide and condom,
    * stable oral/transdermal/injectable hormonal contraceptive regimen without breakthrough uterine bleeding for 2 months prior to Screening visit and a condom used with spermicide,
    * intrauterine device (inserted at least 2 months prior to Screening visit) used with spermicide.

Note: Vasectomy of the partner is not considered sufficient contraception and one of the 4 bulleted methods listed above must be used.

* Agree to use one of the accepted methods of contraception (listed above) during the trial (including the screening period prior to receiving trial medication), and for 1 month after stopping the trial medication.
* Participants enrolled in the placebo arm of Part 1 and who developed akathisia may be eligible for Part 2 in the standard of care arm.

Exclusion Criteria:

* Participants who have a positive screen for drugs with a high potential for abuse. Participants that screen positive for cannabis are permitted.
* Participants who have previously received this compound.
* Participants who are currently participating in another clinical study or have participated in a clinical study within 30 days (except participants enrolled in the Part 1 of the P05145 study).
* Participants who are part of the study staff personnel or family members of the study staff personnel.
* Participants with severe/uncontrolled hypertension will be excluded. Participants with hypertension well controlled on a stable dose of standard antihypertensive medication (excluding beta-blockers) will be eligible.
* Participants with history of coronary artery disease including myocardial infarction (MI), or cerebrovascular disease (stroke, transient ischemic attack [TIA]), or peripheral arterial disease.
* Participants with congestive heart failure or participants with ECGs consistent with ischemic heart disease, sick sinus syndrome or significant Q waves.
* Participants who are found to be at immediate risk of suicide.
* Female participants pregnant or nursing.
* Participants treated by Clozapine will be excluded. A washout period of 6 months prior to dosing will be acceptable for study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-08-15 (Actual); Primary Completion 2008-12-12 (Actual); Study Completion 2009-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Part 1
Arm/Group | Part 1: Preladenant | Part 1: Placebo | Part 2: Preladenant | Part 2: Standard of Care
Started | 19 | 13 | 0 | 0
Completed | 13 | 9 | 0 | 0
Not Completed | 6 | 4 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrew - reason unrelated to treatment | 5 | 2 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Preladenant | Part 1: Placebo | Part 2: Preladenant | Part 2: Standard of Care
Started | 0 | 0 | 8 | 6
Completed | 0 | 0 | 6 | 4
Not Completed | 0 | 0 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrew - reason unrelated to treatment | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Preladenant | Part 1: Placebo | Part 2: Preladenant | Part 2: Standard of Care | Total
Number analyzed (Participants) | 19 | 13 | 8 | 6 | 46
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and <65 years | 19 | 13 | 8 | 6 | 46
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 3 | 2 | 14
  Male | 11 | 12 | 5 | 4 | 32

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Akathisia
Description: Incidence of akathisia is reported as the number of participants who experienced akathisia. Akathisia is defined as a score of 3 on the Barnes akathisia scale (BAS) for 3 consecutive intervals or an akathisia score (BAS) of ≥4 for any single day, or the use of a rescue medication within 13 days of initiating treatment with haloperidol and preladenant. The BAS is scored as follows: objective akathisia, subjective awareness of restlessness and subjective distress related to restlessness are rated on a 4-point scale from 0 - 3 and are summed yielding a total score ranging from 0 (no akathisia) to 9 (severe akathisia).
Time Frame: Up to 13 days
Population: Efficacy analysis population was defined as participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Part 1: Preladenant | Part 1: Placebo
Number analyzed (Participants) | 19 | 13
Participants | 0 | 0

2. Primary Outcome: Part 2: Number of Participants Who Were Treatment Failures
Description: Incidence of treatment failure is reported as the number of participants who were treatment failures. A treatment failure is defined as the failure to achieve at least a 1 point reduction from baseline in BAS score at 24 to 26 hours following study treatment. The BAS is scored as follows: objective akathisia, subjective awareness of restlessness and subjective distress related to restlessness are rated on a 4-point scale from 0 - 3 and are summed yielding a total score ranging from 0 (no akathisia) to 9 (severe akathisia).
Time Frame: Up to 14 days
Population: Efficacy analysis population was defined as participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Part 2: Preladenant | Part 2: Standard of Care
Number analyzed (Participants) | 8 | 6
Participants | 4 | 1

3. Secondary Outcome: Part 1: Mean Global Clinical Impression at Day 14
Description: Global clinical impression (GCI) was administered to assess whether any deterioration is due to akathisia or uncontrolled psychoses. Score on a scale +2 to -2 (+2 represents much improvement, +1 some improvement, 0 no change, -1 some worsening, and -2 much worsening).
Time Frame: Day 14 of Part 1
Population: Efficacy analysis population was defined as participants who received at least one dose of study drug. The study was terminated early by the sponsor due to lack of enrollment. No formal statistical analysis was done due to the very small sample size in this study.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part 1: Preladenant | Part 1: Placebo
Number analyzed (Participants) | 13 | 9
Score on a scale | 0.9231 (0.7596) | 1.7778 (0.4410)

4. Secondary Outcome: Part 1: Mean Positive and Negative Symptom Scale for Schizophrenia (PANSS) Total Score at Day 14
Description: The PANSS is a 30-item clinician-rated instrument for assessing the symptoms of schizophrenia. It consists of 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology subscale (16 items). Positive symptoms refer to an excess or distortion of normal mental status (e.g., delusions). Negative symptoms represent a diminution or loss of normal functions (e.g., emotional withdrawal).
  For each item, symptom severity was rated on a 7-point scale, from 0=absent to 6=extreme. The PANSS total score for each participant was calculated as the sum of the rating assigned to each of the 30 PANSS items, and ranged from 0 to 180 with a higher score indicating greater severity of symptoms. Although the PANSS is traditionally scored with a range of 30-210, with a score of absent = 1 (for each item), for this analysis the range was set from 0-180, with a score of absent = 0 (for each item).
Time Frame: Day 14 of Part 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part 1: Preladenant | Part 1: Placebo
Number analyzed (Participants) | 13 | 9
Score on a scale | 38.4615 (19.4834) | 36.3333 (17.0587)

5. Secondary Outcome: Part 2: Mean GCI at Day 14
Description: The GCI was administered to assess whether any deterioration is due to akathisia or uncontrolled psychoses. Score on a scale +2 to -2 (+2 represents much improvement, +1 some improvement, 0 no change, -1 some worsening, and -2 much worsening).
Time Frame: Day 14 of Part 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part 2: Preladenant | Part 2: Standard of Care
Number analyzed (Participants) | 6 | 4
Score on a scale | 0.6667 (1.0328) | 2.0000 (0.0000)

6. Secondary Outcome: Part 2: PANSS Total Score at Day 14
Description: as for outcome 4
Time Frame: Day 14 of Part 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part 2: Preladenant | Part 2: Standard of Care
Number analyzed (Participants) | 6 | 4
Score on a scale | 43.5000 (28.5430) | 27.75 (11.2361)

ADVERSE EVENTS:
Time Frame: Up to 22 days (including follow-up)
Arm/Group | Part 1: Placebo | Part 1: Preladenant | Part 2: Standard of Care | Part 2: Preladenant
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/19 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 12/13 | 16/19 | 6/6 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=13) | Part 1: Preladenant (N=19) | Part 2: Standard of Care (N=6) | Part 2: Preladenant (N=8)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MALAISE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABSCESS ORAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TINEA PEDIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WEIGHT INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AKATHISIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COGWHEEL RIGIDITY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
DYSKINESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSTONIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1) | 2 (3)
HEAD TITUBATION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (2) | 3 (3) | 2 (3) | 0 (0)
HYPERTONIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OROMANDIBULAR DYSTONIA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
TENSION HEADACHE (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 3 (3) | 1 (2) | 1 (1) | 1 (1)
AFFECTIVE DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PARANOIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCHIZOPHRENIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early by the sponsor due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the study without the prior written consent of the Sponsor. The investigator further agrees to provide to the Sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.